CLINICAL TRIAL: NCT05492591
Title: A Multicenter, Randomized, Active-controlled, Dose-finding Phase II Clinical Study Evaluating the Safety and Efficacy of Peginterferon α1b for Injection in Patients With Herpes Zoster
Brief Title: A Study Exploring Efficacy of Peginterferon in Patients With Herpes Zoster
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIBP-R01
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster; peginterferon; efficacy; safety; postherpetic neuralgia
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, active drug-controlled, dose-finding phase II clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 5 μg/kg of peginterferon α1b for injection in patients with herpes zoster.
  Interventions: Drug: Peginterferon α1b
- Group 2 (Experimental): 6 μg/kg of peginterferon α1b for injection in patients with herpes zoster.
  Interventions: Drug: Peginterferon α1b
- Group 3 (Experimental): 7 μg/kg of peginterferon α1b for injection in patients with herpes zoster.
  Interventions: Drug: Peginterferon α1b
- Group 4 (Experimental): Both valacyclovir tablets and 6 μg/kg of peginterferon α1b for injection plan to be used in patients with herpes zoster.
  Interventions: Drug: Peginterferon α1b with valacyclovir
- Group 5 (Experimental): Both valacyclovir tablets and 7 μg/kg of peginterferon α1b for injection plan to be used in patients with herpes zoster.
  Interventions: Drug: Peginterferon α1b with valacyclovir
- Group 6 (Active Comparator): Only valacyclovir tablets in patients with herpes zoster, positive drug control group.
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Peginterferon α1b — Injecting different doses of the peginterferon α1b into different groups of subjects.
  Arms: Group 1; Group 2; Group 3
Drug: Peginterferon α1b with valacyclovir — Both valacyclovir tablets and different dose of peginterferon α1b plan to be used in different groups of subjects.
  Arms: Group 4; Group 5
Drug: Valacyclovir — Valacyclovir is a positive control drug.
  Arms: Group 6

SUMMARY:
To evaluate the efficacy, optimal dose and efficacy trend of multiple subcutaneous injections of peginterferon α1b in patients with herpes zoster, and provide support for phase III clinical trials.

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, active drug-controlled, dose-finding phase II clinical study. A total of 5 experimental groups and 1 positive drug control group were set up to evaluate the efficacy, optimal dose and efficacy trend of multiple subcutaneous injections of peginterferon α1b in patients with herpes zoster, and provide support for phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give informed consent to the study and agree to participate and give written consent before the study;
* 18 Years to 75 Years （Including 18 and 75 years old），Male or Female;
* Pain VAS score≥3;
* Patients with clinical diagnosis of Herpes Zoster，According to the Chinese Expert Consensus on Herpes zoster (2018) (the rash was asymmetric, unilateral erythematous or maculopapular rash, or clusters of small blisters could appear, and the blister fluid was clear or became cloudy), the appearance of herpes zoster was determined within 3 days (72 hours).

Exclusion Criteria:

* Allergic constitution or history of allergy or known allergy to the test drug product or any component;
* Clinically diagnosed as herpes zoster without rash, disseminated herpes zoster; ear herpes zoster; ocular herpes zoster; with symptoms of viral encephalitis and meningitis; with symptoms of acute gastroenteritis and cystitis; Herpes zoster patients with hemorrhagic, gangrenous clinical manifestations, etc;
* Herpes site with neuralgia caused by other diseases;
* History of serious heart disease, including unstable or uncontrolled angina within 6 months, history of myocardial infarction and other heart disease, epilepsy and other central nervous system disorders, history of autoimmune hepatitis or autoimmune disease, severe liver function Impaired or decompensated cirrhosis, severe mental illness or medical history;
* During the screening period, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 fold ULN;Platelet count <90×109/L;Hemoglobin: male<110g/L，female<100g/L;White blood cell count <3.5×109/L、neutrophil count <1.5×109/L;Renal insufficiency（Cr>1.5 fold ULN and creatinine clearance <60 mL/min），abnormal thyroid function test, positive hepatitis B surface antigen, positive hepatitis C antibody, positive treponema pallidum antibody or positive HIV antibody test in serum virology;
* Previous history of psoriasis;
* Previous organ transplant recipients;
* Patients with active hemorrhagic disease, or severe hematopoietic abnormalities or coagulation disorders within 2 weeks prior to screening;
* Patients with previous history of malignant tumor;
* Patients with a history of severe retinal disease;
* Have received live attenuated vaccine (hepatitis B vaccine, pneumonia vaccine, tetanus vaccine, rabies virus vaccine, cervical cancer vaccine, etc.) within 3 months before screening or planned to receive live attenuated vaccine (hepatitis B vaccine, pneumonia vaccine, tetanus vaccine, rabies virus vaccine, cervical cancer vaccine, etc.) during the trial; have received COVID-19 vaccine within 2 weeks before screening or planned to receive COVID-19 vaccine during the trial;
* Lactating women, blood pregnancy positive subjects (female subjects only), male subjects (or their partners) or female subjects had pregnancy plans or sperm or egg donation plans from 30 days before the study to 3 months after the end of the study and were unwilling to take effective contraceptive measures;
* Participated in any drug or device clinical investigator within 3 months prior to screening;
* Need for driving or precision instrument operation during the study period;
* Within 1 month or 5 half-lives (whichever is the longest) before screening, drugs with therapeutic effect on herpes zoster have been systematically used: interferon, antiviral drugs, immune modulators, glucocorticoids, traditional Chinese medicine/patent medicine, neurotrophic drugs, drugs containing theophylline, etc;
* The patients who had been treated with topical drugs for herpes zoster within 2 weeks before the screening were selected;
* The investigators considered it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Time of stop increasing new blisters/pimples | 5 days after the first dose
  The number of days it took for the herpes to stop increasing (the original blisters/pimples enlarge, and the blisters/pimples increase) after the subjects were screened and enrolled.
Time of target herpes begins to scab | 7 days after the first dose.
  The time taken for the target herpes (where the herpes first occurred when the patient was enrolled) begin to scab after the subjects were screened for enrollment.
Time of complete scabbing of all herpes | 10 days after the first dose.
  The time taken for all the herpes to be completely crusted (the blisters have dried up and crusted) after the subjects were screened and enrolled.

SECONDARY OUTCOMES:
Changes in VAS scores on day 1 from baseline | 1 days after the first dose.
  Changes in VAS scores of subjects on day 1 from baseline.
Changes in VAS scores on day 2 from baseline | 2 days after the first dose.
  Changes in VAS scores of subjects on day 2 from baseline.
Changes in VAS scores on day 3 from baseline | 3 days after the first dose.
  Changes in VAS scores of subjects on day 3 from baseline.
Changes in VAS scores on day 4 from baseline | 4 days after the first dose.
  Changes in VAS scores of subjects on day 4 from baseline.
Changes in VAS scores on day 6 from baseline | 6 days after the first dose.
  Changes in VAS scores of subjects on day 6 from baseline.
Changes in VAS scores on day 10 from baseline | 10 days after the first dose.
  Changes in VAS scores of subjects on day 10 from baseline.
Changes in VAS scores on day 14 from baseline | 14 days after the first dose.
  Changes in VAS scores of subjects on day 14 from baseline.
Changes in VAS scores on day 21 from baseline | 21 days after the first dose.
  Changes in VAS scores of subjects on day 21 from baseline.
Changes in VAS scores on day 27 from baseline | 27 days after the first dose.
  Changes in VAS scores of subjects on day 27 from baseline.
Time that VAS score to drop to ≤2 | 10 days after the first dose.
  The time taken for the VAS score to decrease from baseline ≥3 to ≤2 for the first time after the subjects were screened and enrolled.
Duration time that VAS score to drop to ≤2 | 20 days after the first dose.
  After the subject's VAS score dropped from baseline ≥ 3 to ≤ 2 for the first time, the time that the VAS score remained at ≤ 2.
The time that scabs of blisters fall off | 16 days after the first dose.
  The number of days it took for the scabs of all herpes to completely fall off after the subjects were screened into the group.
Dose of painkiller | 16 days after the first dose.
  The dose of painkiller used within 27 days of the subject's first dose.
Incidence of postherpetic neuralgia | 105 days after the first dose.
  The incidence of hereditary neuralgia within 105 days after the first dose of the subjects. Postherpetic neuralgia is defined as pain lasting one month or more after the rash has healed (ie, complete exfoliation).

OTHER OUTCOMES:
Postherpetic neuralgia duration | 105 days after the first dose.
  The duration of postherpetic neuralgia within 105 days after the subject's first dose.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences Dermatology Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No